CLINICAL TRIAL: NCT00106522
Title: A Randomized, Double-blind Study of Safety and Reduction in Signs and Symptoms During Treatment With Tocilizumab Versus Placebo, in Combination With Methotrexate, in Patients With Moderate to Severe Active Rheumatoid Arthritis and Inadequate Response to Anti-TNF Therapy
Brief Title: A Study to Assess the Effect of Tocilizumab + Methotrexate on Signs and Symptoms in Patients With Moderate to Severe Active Rheumatoid Arthritis Currently on Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA18062
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- 2 (Experimental)
  Interventions: Drug: Methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- 3 (Placebo Comparator)
  Interventions: Drug: Methotrexate; Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — 10-25mg weekly
Drug: Placebo — iv every 4 weeks
  Arms: 3
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks
  Arms: 2
Drug: tocilizumab [RoActemra/Actemra] — 4mg/kg iv every 4 weeks
  Arms: 1

SUMMARY:
This 3 arm study will compare the safety and efficacy, with regard to reduction of signs and symptoms, of tocilizumab versus placebo in combination with methotrexate (MTX) in patients with moderate to severe active rheumatoid arthritis (RA) currently on MTX therapy, and who have had an inadequate response to prior therapy with an anti-tumor necrosis factor (anti-TNF) agent. Patients will be randomized to receive tocilizumab 4mg/kg iv, tocilizumab 8mg/kg or placebo iv, every 4 weeks. All patients will also receive methotrexate 10-25mg/week. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age with moderate to severe active RA for at least 6 months;
* inadequate response to current anti-rheumatic therapies, including MTX;
* inadequate response or intolerance to treatment with 1 or more anti-TNF therapies within 1 year of entering study;
* on stable MTX for at least 8 weeks before entering study;
* patients of reproductive potential must be using reliable methods of contraception.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks before screening, or planned major surgery within 6 months after entering study;
* women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 24
AEs, laboratory parameters, vital signs, ECGs. | Throughout study

SECONDARY OUTCOMES:
Percentage of patients with ACR 50 and ACR 70 responses | Week 24
Mean changes in parameters of ACR core set | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (151):
- United States (84):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Fullerton, California
  - Long Beach, California
  - Los Angeles, California
  - Palm Desert, California
  - San Diego, California
  - Santa Maria, California
  - Torrance, California
  - Colorado Springs, Colorado
  - Aventura, Florida
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Palm Habor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Tavares, Florida
  - West Palm Beach, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Bowling Green, Kentucky
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Wheaton, Maryland
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Duluth, Minnesota
  - Rochester, Minnesota
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Billings, Montana
  - Missoula, Montana
  - Las Vegas, Nevada
  - Medford, New Jersey
  - Mercerville, New Jersey
  - Teaneck, New Jersey
  - Albany, New York
  - Binghamton, New York
  - Great Neck, New York
  - Johnson City, New York
  - New York, New York
  - Orchard Park, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Bismarck, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Danville, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Willow Grove, Pennsylvania
  - Hickory Grove, South Carolina
  - Jackson, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Ogden, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Salem, Virginia
  - Seattle, Washington
  - Glendale, Wisconsin
- Australia (4):
  - Malvern
  - Shenton Park
  - Sydney
  - Woolloongabba
- Belgium (3):
  - Aalst
  - Hasselt
  - Merksem
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Burlington, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (9):
  - Amiens
  - Bordeaux
  - Le Kremlin-Bicêtre
  - Lille
  - Lyon
  - Nice
  - Paris
  - Strasbourg
  - Toulouse
- Germany (8):
  - Berlin
  - Cologne
  - Dresden
  - Gommern
  - Herne
  - München
  - Wiesbaden
  - Würzburg
- Reykjavik, Iceland
- Italy (6):
  - Brescia
  - Milan
  - Padua
  - Pavia
  - Pisa
  - Udine
- Guadalajara, Mexico
- Netherlands (2):
  - Enschede
  - Nijmegen
- Ponce, Puerto Rico
- Sweden (4):
  - Jönköping
  - Karlstad
  - Malmo
  - Stockholm
- Lausanne, Switzerland
- United Kingdom (17):
  - Basingstoke
  - Bath
  - Birmingham
  - Cannock
  - Derby
  - Lancaster
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Middlesbrough
  - Newcastle upon Tyne
  - Norwich
  - Oxford
  - Salford
  - Southampton
  - Stoke-on-Trent

REFERENCES:
- [Derived] Vieira MC, Zwillich SH, Jansen JP, Smiechowski B, Spurden D, Wallenstein GV. Tofacitinib Versus Biologic Treatments in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Tumor Necrosis Factor Inhibitors: Results From a Network Meta-analysis. Clin Ther. 2016 Dec;38(12):2628-2641.e5. doi: 10.1016/j.clinthera.2016.11.004. Epub 2016 Nov 24. PMID 27889300
- [Derived] Keystone EC, Anisfeld A, Ogale S, Devenport JN, Curtis JR. Continued benefit of tocilizumab plus disease-modifying antirheumatic drug therapy in patients with rheumatoid arthritis and inadequate clinical responses by week 8 of treatment. J Rheumatol. 2014 Feb;41(2):216-26. doi: 10.3899/jrheum.130489. Epub 2014 Jan 15. PMID 24429164
- [Derived] Strand V, Burmester GR, Ogale S, Devenport J, John A, Emery P. Improvements in health-related quality of life after treatment with tocilizumab in patients with rheumatoid arthritis refractory to tumour necrosis factor inhibitors: results from the 24-week randomized controlled RADIATE study. Rheumatology (Oxford). 2012 Oct;51(10):1860-9. doi: 10.1093/rheumatology/kes131. Epub 2012 Jun 28. PMID 22753773
- [Derived] Karsdal MA, Schett G, Emery P, Harari O, Byrjalsen I, Kenwright A, Bay-Jensen AC, Platt A. IL-6 receptor inhibition positively modulates bone balance in rheumatoid arthritis patients with an inadequate response to anti-tumor necrosis factor therapy: biochemical marker analysis of bone metabolism in the tocilizumab RADIATE study (NCT00106522). Semin Arthritis Rheum. 2012 Oct;42(2):131-9. doi: 10.1016/j.semarthrit.2012.01.004. Epub 2012 Mar 6. PMID 22397953
- [Derived] Emery P, Keystone E, Tony HP, Cantagrel A, van Vollenhoven R, Sanchez A, Alecock E, Lee J, Kremer J. IL-6 receptor inhibition with tocilizumab improves treatment outcomes in patients with rheumatoid arthritis refractory to anti-tumour necrosis factor biologicals: results from a 24-week multicentre randomised placebo-controlled trial. Ann Rheum Dis. 2008 Nov;67(11):1516-23. doi: 10.1136/ard.2008.092932. Epub 2008 Jul 14. PMID 18625622